CLINICAL TRIAL: NCT00158522
Title: Clinical Trial of the Efficacy of Pegylated Interferon (PEG-IFNα-2a) Alone in Egyptian Patients With Acute Hepatitis C
Brief Title: Efficacy of Pegylated Interferon Alone in Egyptian Patients With Acute Hepatitis C (ANRS 1213)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Director, ANRS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 1213
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-02

CONDITIONS: Hepatitis C
Keywords: Acute hepatitis C; Genotype 4; Pegylated Interferon; Egypt
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: pegylated interferon alpha2a

INTERVENTIONS:
Drug: pegylated interferon alpha2a

SUMMARY:
Acute hepatitis C is a liver disease related to a virus: hepatitis C virus (HCV). The type of Hepatitis C Virus present in Egypt (genotype 4), has the reputation to respond poorly to treatment at the chronic hepatitis stage. Without treatment, 85% of patients with acute hepatitis C become chronically HCV infected which means that the virus stays present in the body. Pegylated Interferon is a new form of Interferon that stays in the body for longer time and allows the patient to take less injection per week. It has also proved to be more effective than standard Interferon in treatment of chronic hepatitis C.

DETAILED DESCRIPTION:
Egypt is the country with the highest HCV prevalence worldwide, and the number of infected Egyptians is estimated around 8 million. HCV incidence is high as well, and a typical hepatology department in Cairo diagnoses between 5 and 10 acute hepatitis C per month. The HCV genotype circulating in Egypt is genotype 4. This genotype has the reputation to respond poorly to treatment at the chronic hepatitis stage. It would therefore be interesting to assess the treatment efficacy at the acute stage. This study will evaluate the efficacy of pegylated interferon (peg-IFNα-2a) alone in Egyptian patients with acute hepatitis C.

The study primary objective is to evaluate the efficacy and tolerance of pegylated interferon (peg-IFNα-2a) alone in Egyptian patients with acute hepatitis C.

Methods: One arm clinical trial. Follow-up duration: 36 to 48 weeks depending on response to treatment.

Main inclusion criteria: ALT> 3*N; HCV RNA positive by PCR and negative HCV serology at first presentation or positive HCV serology with a clear and unique exposure within 2 months prior the acute hepatitis episode; no prior treatment with IFNα, peg-IFNα and ribavirin; signed informed consent.

Main exclusion criteria : Liver disease other than hepatitis C. Treatment strategy: Peg-IFNα-2a 180microg/week (subcutaneous injection) for 12 weeks. Patients with positive HCV RNA by qualitative PCR at the end of the 12 weeks treatment period will be offered to continue on the same regimen up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Acute hepatitis C:(1)ALT over 3x normal values ; IgM anti-HAV, IgM anti-HBc negative antibody ; negative HCV antibodies (3rd generation ELISA) and positive HCV PCR at first presentation, or, (2)ALT over 4x normal values ; IgM anti-HAV, IgM anti-HBc, CMV, EBV and toxoplasmoses negative antibody and negative HEV PCR ; Positive HCV antibodies (3rd generation ELISA) and positive HCV PCR at first presentation ; a clear history of exposure within 2 months prior the time of diagnosis ; no exposure to hepatotoxic drug or pesticide within 2 weeks prior the time of diagnosis
* Patients without chronic liver disease
* HBsAg negative
* Hemoglobin over or equal to 11g/dl
* Leucocytes over or equal to 3000/mm3
* Polynuclear neutrophils over or equal to 1500/mm3
* Platelets over or equal to 100 000/mm3
* Blood creatinin less or equal to 150 micromol/l
* Blood uric acid within the normal limits of the investigating center
* Normal TSH
* Antinuclear antibodies < 1/160
* Fasting blood sugar 70-115 mg/dl ; if glucose intolerance or diabetes, HbA1C less or equal to 8,5%
* Normal ophthalmologic examination for all patients
* Effective contraception during the treatment period.
* No breastfeeding during the study period
* Signed informed consent

Exclusion Criteria:

* Co-infection with hepatitis B (positive HBs antigen)
* Hemochromatosis
* Alpha-1 anti-trypsin deficiency
* Wilson disease
* Alcoholism-related liver disease
* Gilbert disease
* Liver cirrhosis
* Hepatocellular carcinoma.
* Alcohol intake over 50g/day for males and 40 g/day for females
* Intravenous drug use
* Psychiatric disease: history of severe nervous breakdown or severe psychiatric diseases such as major psychosis, suicidal ideas, suicide attempts…
* Epilepsy
* Auto-immune disease
* Heart disease in the six months preceding enrolment - patients with significant changes at EKG
* Uncontrolled diabetes
* Chronic respiratory insufficiency with hypoxemia under 10 kPa
* Medical or surgical condition non-stabilized, with life expectancy lower than two years
* Pregnancy or breastfeeding
* Unavailability for regular follow-up during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Disappearance of HCV RNA by qualitative PCR 24 weeks after the end of treatment

SECONDARY OUTCOMES:
Changes in HCV RNA load
Normalization of ALT during treatment and 24 weeks after the end of treatment
Study of side effects

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa K Mohamed, Principal Investigator — National Hepatology and Tropical Medicine Research Institute; Fontanet Arnaud, Study Chair — Institut Pasteur de Paris
Locations (1):
- National Hepatology and Tropical Medicine Research Institute, Cairo, Egypt

REFERENCES:
- [Background] Bakr I, Rekacewicz C, El Hosseiny M, Ismail S, El Daly M, El-Kafrawy S, Esmat G, Hamid MA, Mohamed MK, Fontanet A. Higher clearance of hepatitis C virus infection in females compared with males. Gut. 2006 Aug;55(8):1183-7. doi: 10.1136/gut.2005.078147. Epub 2006 Jan 24. PMID 16434426
- [Background] El Gaafary MM, Rekacewicz C, Abdel-Rahman AG, Allam MF, El Hosseiny M, Hamid MA, Colombani F, Sultan Y, El-Aidy S, Fontanet A, Mohamed MK. Surveillance of acute hepatitis C in Cairo, Egypt. J Med Virol. 2005 Aug;76(4):520-5. doi: 10.1002/jmv.20392. PMID 15977225
- See also: Sponsor web page - information in french and english — http://www.anrs.fr